CLINICAL TRIAL: NCT01636648
Title: Enable I Long-term Follow-up Study
Status: Terminated | Type: Observational
Why Stopped: Device was sunset from the market in May2015. No longer need for long term data.
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: En_2012
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Insufficiency
Keywords: Aortic Valve Replacement; Aortic Valve Bioprosthesis
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Aortic Valve Replacement — Aortic Valve Replacement with Medtronic ATS 3f ENABLE® Aortic Bioprosthesis Model 6000

SUMMARY:
This was a prospective, non-randomized, multi-center, non-interventional post-market study. The study was a post-market long-term follow-up study based on the same cohort of patients (148 patients) enrolled in a previous investigational study from March 2007 to December 2009 (ATS 3f Enable™ Aortic Bioprosthesis Model 6000, number S2005) involving 10 European sites. Patient follow-up took place on a yearly basis up to 10 years after the implant/enrollment. The primary objective of this study was to evaluate the safety and effectiveness of the Medtronic ATS Enable Aortic Bioprosthesis during long-term follow-up.

As this was an observational study, safety and efficacy data were summarized and described. There was no statistically powered study hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were enrolled and implanted for the ATS 3f Enable™ Aortic Bioprosthesis Model 6000, number S2005
* Patient willing to sign the new Data Release form (DRF) or Patient Informed Consent (PIC) for the post-market study (what is applicable for the study due to local requirements and regulations)

Exclusion Criteria:

* ATS 3f Enable™ Aortic Bioprosthesis Model 6000 was explanted
* Patient died
* Patient lost to follow-up
* Patient withdrew consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were enrolled and implanted during the previous investigational study named "ATS 3f Enable™ Aortic Bioprosthesis Model 6000" (study number S2005).
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2012-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Assess the Long-term safety of the Medtronic ATS Enable Aortic Bioprosthesis | 10 Years Post-Procedure
  Long-term safety will be assessed by collecting following reported adverse events addressed: Migration, Valve Related Thromboembolism, Valvular thrombosis, Haemorrhage, Perivalvular Leak, Endocarditis, Hmolysis, Structural valve Deterioration, Non-Structural Dysfunction, Reoperation, Explant and Death.
Assess the Long-term Clinical Effectiveness of the Medtronic ATS Enable Aortic Bioprosthesis: NYHA Functional Classification | 10 Years Post-Procedure
  Long-term clinical effectiveness of the Aortic Bioprosthesis will be assessed by collecting the NYHA-class of enrolled subjects over a period of time, following surgery.
Long-term Effectiveness of the Medtronic ATS Enable Aortic Bioprosthesis: Hemodynamic Performance | 10 Years Post-Procedure
  Hemodynamic performance of the Aortic Bioprosthesis will be assessed by specific echocardiography measurements

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Carrel, Prof., Principal Investigator — Inselspital Bern, Klinik für Herz-und Gefasschirurgie, CH-3010 Bern
Locations (6):
- Germany (3):
  - Johann Wolfgang Goethe University, Frankfurt
  - University Medical Center Freiburg, Freiburg im Breisgau
  - University Medical Center Kiel, Kiel
- Jagellonian University, John Paul the II Hospital, Krakow, Poland
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martens S, Sadowski J, Eckstein FS, Bartus K, Kapelak B, Sievers HH, Schlensak C, Carrel T. Clinical experience with the ATS 3f Enable(R) Sutureless Bioprosthesis. Eur J Cardiothorac Surg. 2011 Sep;40(3):749-55. doi: 10.1016/j.ejcts.2010.12.068. Epub 2011 Feb 20. PMID 21342776
- [Background] Englberger L, Carrel TP, Doss M, Sadowski J, Bartus K, Eckstein FF, Asch FM, Martens S. Clinical performance of a sutureless aortic bioprosthesis: five-year results of the 3f Enable long-term follow-up study. J Thorac Cardiovasc Surg. 2014 Oct;148(4):1681-7. doi: 10.1016/j.jtcvs.2014.03.054. Epub 2014 Apr 4. PMID 24787699